CLINICAL TRIAL: NCT02844946
Title: One-Day Life Skills Workshop for Veterans With TBI, Pain and Psychopathology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: D2209-P
Record Dates: First submitted 2016-07-22; First posted 2016-07-26 (Estimated); Results first posted 2019-08-28 (Actual); Last update posted 2021-12-02 (Actual); Status verified 2021-11

CONDITIONS: Mild Traumatic Brain Injury; Distress-based Psychopathology; Chronic Pain
Keywords: Acceptance and Commitment Therapy; mild Traumatic Brain Injury; Veterans; Post Traumatic Stress Disorder
MeSH Terms: conditions — Brain Concussion; Chronic Pain; Stress Disorders, Post-Traumatic | interventions — Acceptance and Commitment Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ACT on Life (Experimental): One day workshop aimed at providing Veterans with new tools and skills needed to pursue valued goals and directions in the face of life's challenges. Mindfulness, acceptance, values clarification, and goal-setting will be taught.
  Interventions: Behavioral: Acceptance and Commitment Therapy
- Treatment as Usual (No Intervention): Veterans will continue receiving care as usual.

INTERVENTIONS:
Behavioral: Acceptance and Commitment Therapy — Contextually focused form of cognitive behavioral psychotherapy that uses MINDFULNESS and behavioral activation to increase patients' psychological flexibility in areas such as ability to engage in values-based, positive behaviors while experiencing difficult thoughts, emotions, or sensations.
  Arms: ACT on Life

SUMMARY:
Traumatic brain injury (TBI) is the signature wound of Veterans returning from the recent operations in Iraq and Afghanistan (i.e OIF/OEF/OND), with up to 20 percent experiencing persistent post-concussive symptoms. Among Veterans with mild TBI, the majority also experience significant distress, including depression and post-traumatic stress disorder, as well as persistent pain. Importantly, significant stigma is associated with seeking mental health care among Veterans; and poor management of multiple conditions results in increased morbidity and mortality, increased risk for suicide, and significantly decreased quality of life. Thus the challenge for treatment providers is to provide a unified and acceptable intervention for Veterans with these interdependent systemic comorbid concerns. The aim of this proposal is to develop, refine, and evaluate a 1-day trans-diagnostic (i.e., applies to more than one diagnosis) "life skills workshop" to help Veterans develop skills needed to pursue valued goals in the face of life's challenges.

DETAILED DESCRIPTION:
Traumatic brain injury (TBI) is the signature wound of Veterans returning from Operations Iraqi Freedom, Enduring Freedom and Operation New Dawn (OIF/OEF/OND), with up to 20 percent experiencing persistent post-concussive symptoms. Among those with a mild TBI (mTBI) diagnosis, the majority also suffers from stress-based psychopathology, including depression, post-traumatic stress disorder, and other anxiety disorders, as well as persistent pain. Poor management of multiple conditions results in increased morbidity and mortality, increased risk for suicide, and significantly decreased quality of life. Importantly, the association between seeking mental health care and stigma among Veterans is high. Veterans are often unwilling to seek mental health services due to concern that receiving such care would negatively impact their careers and the belief that they should be able to overcome psychological difficulties on their own. Furthermore availability of specialty services is limited for Veterans living in rural settings. Thus the challenge for treatment providers is to provide a unified, efficient, accessible, and acceptable intervention for Veterans with these interdependent systemic comorbid concerns. Acceptance and Commitment Therapy (ACT) is a trans-diagnostic (i.e., applies to more than one diagnosis) behavioral intervention aimed at helping individuals develop the skills needed to pursue valued goals and directions in the face of life's challenges. It provides a unified model of behavior change that has shown promise in treating depression and anxiety, as well as chronic medical conditions. Importantly, ACT has been effectively implemented in various treatment-delivery formats, including 1-day workshops. This flexibility in delivery format allows focus to be placed on how best to package and deliver the intervention to meet the needs of this Veteran patient population, to ensure treatment adherence, and also to increase chances of dissemination into clinical settings. Providing a 1-day ACT "workshop" for Veterans with mTBI, pain, and mental health problems will allow unitary comprehensive care for the range of emotional, physical, and cognitive symptoms experienced by these Veterans. Presenting the treatment as a "workshop" rather than "therapy" will also be better suited for the Veterans who may not be explicitly seeking specialized mental health care. Finally, a 1-day workshop ensures treatment adherence and completion, the lack of which is often the greatest obstacle to effective delivery of mental health services.

The aims of this study are to:

1. develop a 1-day (5-hour) "ACT on Life" workshop tailored specifically for Veterans with mTBI, stress-based psychopathology, and pain; a multi-disciplinary team of a clinical psychologist, neuropsychiatrist, cognitive psychologist, and anthropologist will provide expert input for use in producing the therapist intervention and patient manual;
2. enroll 10 Veterans with mTBI, stress-based psychopathology, and pain in the "ACT on Life" workshop to obtain qualitative and quantitative feedback from Veterans about the intervention; use Veteran feedback to refine the treatment procedures and manuals; and examine feasibility and acceptability of the intervention; (this is called Pilot 1 and is the first time we recruited participants to obtain feedback on the intervention); and 3) randomize 30 Veterans with mTBI, pain, and stress-based psychopathology to the refined "ACT on Life" workshop or to Treatment as usual (TAU) to examine the preliminary efficacy of the intervention on quality of life and functioning, stress-based symptoms of psychopathology, and pain interference (this is called Pilot 2 and quantitative feedback was obtained). The results section will reflect data from Pilot 2.

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years of age
* Clinically significant psychological distress as operationalized by a diagnosis of major depressive disorder, generalized anxiety disorder, or PTSD
* Life time history of Mild TBI

  * the Department of Veterans Affairs and the Department of Defense define TBI as a traumatically induced structural injury and/or physiological disruption of brain function that is associated with any period of loss of or a decreased level of consciousness
  * any loss of memory for events immediately before or after the injury
  * any alteration in mental state at the time of the injury
  * neurological deficits that may or may not be transient
  * or an intracranial lesion
* Mild TBI is characterized by loss of consciousness less than 30 minutes, a period of post-traumatic amnesia less than 24 hours or, if available, a Glasgow Coma Scale score of 13 to 15
* Presence in medical chart of chronic pain including headache, musculoskeletal pain or neuropathic pain
* Stable dose of psychiatric medications for the past 8 weeks

Exclusion Criteria:

* History of primary psychotic disorder, e.g.,:

  * schizophrenia
  * schizoaffective disorder
* A diagnosis of substance dependence in the year prior to enrollment in the study
* Active suicidal ideation
* Homicidal ideation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2016-10-03 (Actual); Primary Completion 2018-09-03 (Actual); Study Completion 2018-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lilian N. Dindo, PhD, Principal Investigator — Michael E. DeBakey VA Medical Center, Houston, TX
Locations (1):
- Michael E. DeBakey VA Medical Center, Houston, TX, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Dindo L, Johnson AL, Lang B, Rodrigues M, Martin L, Jorge R. Development and evaluation of an 1-day Acceptance and Commitment Therapy workshop for Veterans with comorbid chronic pain, TBI, and psychological distress: Outcomes from a pilot study. Contemp Clin Trials. 2020 Mar;90:105954. doi: 10.1016/j.cct.2020.105954. Epub 2020 Feb 4. PMID 32032736

RESULTS

PARTICIPANT FLOW:
Groups:
- ACT on Life: One day workshop aimed at providing Veterans with new tools and skills needed to pursue valued goals and directions in the face of life?s challenges. Mindfulness, acceptance, values clarification, and goal-setting will be taught.
  Acceptance and Commitment Therapy: Contextually focused form of cognitive behavioral psychotherapy that uses MINDFULNESS and behavioral activation to increase patients' psychological flexibility in areas such as ability to engage in values-based, positive behaviors while experiencing difficult thoughts, emotions, or sensations.
Period: Overall Study
Arm/Group | ACT on Life | Treatment as Usual
Started | 27 | 12
Completed | 20 | 12
Not Completed | 7 | 0
Not completed — Lost to Follow-up | 7 | 0

BASELINE CHARACTERISTICS:
Population: Of note, initially 27 participants were assigned to the ACT on Life Condition. However, only 19 of those were eligible, with valid data, and actually began the workshop.
Groups:
- Total: Total of all reporting groups
Arm/Group | ACT on Life | Treatment as Usual | Total
Number analyzed (Participants) | 19 | 12 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.7 (6.3) | 34.7 (5.8) | 37.2 (6.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 19 | 12 | 31
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 8 | 5 | 13
  African American | 4 | 2 | 6
  Hispanic/Latino | 4 | 3 | 7
  Other | 3 | 2 | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 19 | 12 | 31
World Health Organization-Quality of Life (WHO-QOL) [Mean (Standard Deviation); unit: units on a scale] — The general Quality of Life scale includes 2 items that measure overall QOL and general health. Items scored are scored from 1-5 so the range for the this scale is 2-10 with higher scores representing higher quality of life.
  units on a scale | 6.11 (1.97) | 5.17 (1.90) | 5.7 (1.9)
The Depression Anxiety and Stress Scale (DASS-21) [Mean (Standard Deviation); unit: units on a scale] — This 21-item measure consists of three self-report scales that measure current symptoms of depression, anxiety, and stress and a total score. It has been used extensively in clinical trials, including those with military populations. Higher scores represent greater distress and scores range from 0-126.
  units on a scale | 53.4 (6.3) | 59.7 (8.0) | 55.1 (7.2)
The Brief Pain Inventory (BPI) Severity [Mean (Standard Deviation); unit: units on a scale] — The BPI severity scale assesses pain at its "worst," "least," "average," and "now" (current pain). A composite of the four pain items (a mean severity score) is used here as recommended for assessing pain in clinical trials. Higher scores represent greater severity (0-10).
  units on a scale | 5.5 (.4) | 4.5 (.5) | 5.0 (.4)
World Health Organization Disability Assessment Schedule II (WHODAS-II) [Mean (Standard Deviation); unit: units on a scale] — This is a self-report measure that assesses behavioral and functional impairments as a separate domain from disease symptoms. Higher scores indicate higher disability (from 0-100).
  units on a scale | 40.9 (5.2) | 40.8 (7.1) | 40.9 (6)
Military to Civilian Questionnaire (M2C-Q) [Mean (Standard Deviation); unit: units on a scale] — This 16-item self-report measure assesses post-deployment difficulties with reintegration during the previous month. Respondents rate the level of difficulty on a 5-point scale from No Difficulty to Extreme Difficulty (0-4). The following domains are covered by the M2C-Q: Social relations, community engagement, perceived meaning in life, self-care and leisure, and parenting. The total score is the average of the 16 items. Higher scores reflecting greater difficulty with reintegration.
  units on a scale | 2.0 (.21) | 2.0 (.27) | 2.0 (.23)
PTSD Checklist-Civilian Version (PCL-C) [Mean (Standard Deviation); unit: units on a scale] — PCL-C is a 17-item self-report questionnaire assessing the presence and severity of DSM-IV symptoms of PTSD during the past month. All items are added for a total severity score. Higher scores represent greater severity of PTSD symptoms. Scores range from 1-85.
  units on a scale | 56.3 (4.3) | 56.2 (5.4) | 56.2 (4.6)
Acceptance and Action Questionnaire-II (AAQ-II) [Mean (Standard Deviation); unit: units on a scale] — The AAQ-II is an ACT-specific self-report measure of psychological inflexibility. Seven items are rated on a 7-point scale, ranging from 1 ("never true") to 7 ("always true"), with higher scores reflecting greater inflexibility. Scores range from 1-49.
  units on a scale | 27.3 (2.8) | 29.5 (3.7) | 28.4 (3.2)

OUTCOME MEASURES:

1. Primary Outcome: World Health Organization-Quality of Life (WHO-QOL)
Description: Quality of Life. The general Quality of Life scale includes 2 items that measure overall QOL and general health. Items scored are scored from 1-5 so the range for the this scale is 2-10 with higher scores representing higher quality of life.
Time Frame: Through study completion, an average of 3 months following workshop attendance
Population: 27 participants were assigned to the ACT on Life Condition. Only 19 were eligible, with valid data, and actually began the workshop.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | ACT on Life | Treatment as Usual
Number analyzed (Participants) | 19 | 12
units on a scale | 6.11 (1.94) | 5.20 (1.55)

2. Primary Outcome: Depression Anxiety and Stress Scale (DASS-21)
Description: Consists of three self-report scales that measure current depression, anxiety, and stress. This 21-item measure consists of three self-report scales that measure current symptoms of depression, anxiety, and stress and a total score. It has been used extensively in clinical trials, including those with military populations. Higher scores represent greater distress and scores range from 0-126.
Time Frame: Through study completion, an average of 3 months following workshop attendance
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | ACT on Life | Treatment as Usual
Number analyzed (Participants) | 19 | 12
units on a scale | 42.7 (6.3) | 65.6 (8.3)

3. Primary Outcome: Brief Pain Inventory (BPI)
Description: Assesses the severity of pain and the impact of pain on daily functions. The BPI severity scale assesses pain at its "worst," "least," "average," and "now" (current pain). A composite of the four pain items (a mean severity score) is used here as recommended for assessing pain in clinical trials. Higher scores represent greater severity (0-10).
Time Frame: Through study completion, an average of 3 months following workshop attendance
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ACT on Life | Treatment as Usual
Number analyzed (Participants) | 19 | 12
units on a scale | 5.3 (.5) | 4.2 (.7)

4. Primary Outcome: World Health Organization Disability Assessment Schedule II (WHODAS-II)
Description: Assesses functioning and disability due to health conditions. Six domains are covered: understanding and communicating, getting around, self-care, getting along with people, life act. This is a self-report measure that assesses behavioral and functional impairments as a separate domain from disease symptoms. Higher scores indicate higher disability (from 0-100).
Time Frame: Through study completion, an average of 3 months following workshop attendance
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | ACT on Life | Treatment as Usual
Number analyzed (Participants) | 19 | 12
units on a scale | 38.3 (5.6) | 41.7 (7.7)

5. Secondary Outcome: Military to Civilian Questionnaire (M2C-Q)
Description: This 16-item self-report measure assesses post-deployment difficulties with reintegration during the previous month. Respondents rate the level of difficulty on a 5-point scale from No Difficulty to Extreme Difficulty (0-4). The following domains are covered by the M2C-Q: Social relations, community engagement, perceived meaning in life, self-care and leisure, and parenting. The total score is the average of the 16 items. Higher scores reflecting greater difficulty with reintegration.
Time Frame: Through study completion, an average of 3 months following workshop attendance
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | ACT on Life | Treatment as Usual
Number analyzed (Participants) | 19 | 12
units on a scale | 1.81 (.22) | 2.14 (.30)

6. Secondary Outcome: PTSD Checklist-Civilian Version (PCL-C)
Description: PCL-C is a 17-item self-report questionnaire assessing the presence and severity of DSM-IV symptoms of PTSD during the past month. All items are added for a total severity score. Higher scores represent greater severity of PTSD symptoms. Scores range from 1-85.
Time Frame: Through study completion, an average of 3 months following workshop attendance
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | ACT on Life | Treatment as Usual
Number analyzed (Participants) | 19 | 12
units on a scale | 49.2 (3.8) | 54.4 (4.8)

7. Secondary Outcome: Acceptance and Action Questionnaire-II (AAQ-II)
Description: The AAQ-II is an ACT-specific self-report measure of psychological inflexibility. Seven items are rated on a 7-point scale, ranging from 1 ("never true") to 7 ("always true"), with higher scores reflecting greater inflexibility. Scores range from 1-49. Example items include, "Emotions cause problems in my life," and "My painful memories prevent me from having a fulfilling life." It has been shown to have good internal consistency and validity and also to mediate behavioral outcomes in ACT interventions.
Time Frame: Through study completion, an average of 3 months following workshop attendance
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | ACT on Life | Treatment as Usual
Number analyzed (Participants) | 19 | 12
units on a scale | 22.8 (2.8) | 30.3 (3.8)

ADVERSE EVENTS:
Time Frame: Through study completion, up to 3 months following workshop attendance.
Description: This is a low-risk study. The investigators are simply providing a workshop to Veterans to teach them more about their difficulties and new ways they may cope. However, if at any time during the study we obtained information about significant and imminent suicidality, we would follow-up by doing a suicide risk assessment and making immediate referrals.
Arm/Group | ACT on Life | Treatment as Usual
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/12
Other Adverse Events (participants affected / at risk) | 0/19 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-19): https://cdn.clinicaltrials.gov/large-docs/46/NCT02844946/Prot_SAP_000.pdf